CLINICAL TRIAL: NCT03850132
Title: The Effect of Receiving a FAM-SOTC Intervention Before and in the Bereavement Phase (FAM-SOTC-PL) on Bereaved Family Cancer Caregivers Outcomes: A Quasi-experimental Study
Brief Title: Family Cancer Caregivers Receiving a Specific Supportive Care Intervention Pre- and Postloss
Acronym: FAM-SOTC-PL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UIceland-12018
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-12

CONDITIONS: Bereavement
Keywords: Caregivers; Cancer; Palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAM-SOTC-PL (Experimental): Grief responses, levels of vulnerability, measured using the Adult Attitude to Grief scale (AAG), a self-administered questionnaire
  Interventions: Behavioral: FAM-SOTC-PL

INTERVENTIONS:
Behavioral: FAM-SOTC-PL — The adapted FAM-SOTC-PL intervention was delivered at the home of the participants and focuses on supporting the effective, cognitive, and behavioural domains of the bereaved family caregivers experience by targeting concerns/issues in these categories. The FAM-SOTC-PL comprises of the following five components:
  1. Drawing forward narratives about the pre- and post-loss experience.
  2. Asking therapeutic/interventive questions, emphasising on the most pressing concerns also assessing health issues.
  3. Validating/acknowledging emotional responses.
  4. Assessing the need for specific information and recommendations regarding bereavement.
  5. The use of commendation/commending strengths, by focusing on and affirming the strengths of the family caregiver.

SUMMARY:
Background and study aims The effect of cancer caregiving may have profound impact on the psychosocial health of family caregivers and become evident after loss. Grief following the loss of a close relative is one of the most emotional challenging experience faced by family caregivers. Providing a family based intervention before and after a close relatives´death may positively impact bereavement outcomes. This study aims to assess the impact of a continuing specific supportive care intervention on bereaved family caregivers grief response scores and psychological distress following the loss of a close relative when offered before and after death because of cancer.

DETAILED DESCRIPTION:
This clinical trial is part of a broader research study (registered trial intervention ISRCTN21786830) which aimed to evaluate a palliative care nurse-led family-oriented intervention Family-Strengths Oriented Therapeutic Conversation (FAM-SOTC) to support family caregivers of a close relative with advanced/final stage cancer, in the context of the family when receiving specialized palliative home-care. The purpose of the current trial is to investigate the effects of the FAM-SOTC intervention when additionally delivering the third session of the intervention in this trial; an adapted version; FAM-SOTC Post-Loss and repeated post-intervention measures at 3, 5 and six months post-loss completed by bereaved family caregivers who have prior participated in the FAM-SOTC trial intervention pre-loss are compared to measures at 3, 5 and six months post-loss among bereaved family caregivers in a control group who received usual care pre- and post-loss from the palliative home-care unit. The FAM-SOTC intervention and the FAM-SOTC Post Loss intervention is delivered simultaneously in two separate clinical trials, where two sessions were delivered pre-loss (FAM-SOTC) and one session delivered post-loss (FAM-SOTC-PL).

ELIGIBILITY:
Inclusion Criteria:

* The eligibility criteria is that the primary family caregivers (who had been identified by the patient pre-death) are aged 18 years or older, bereaved due to cancer and that three months have passed since the deceased has died. Additional inclusion criteria is that the family caregivers have received care from a specialised palliative home-care unit at a university hospital in the advanced and final stage of their close relatives´ cancer trajectory.

Exclusion Criteria:

* Non cancer and not being participating in another family level psycho-social intervention research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-07-27 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Change in Depression | 3, 5, and 6 months
  The Depression Anxiety Stress Scale - DASS (Lovibond & Lovibond, 1995) is used. The DASS is a 42-item self-report instrument with 3 sub-scales. Each scale comprises 14 items assessing the negative emotional states of depression, anxiety and stress.
Change in Anxiety | 3, 5, and 6 months
  The Depression Anxiety Stress Scale - DASS (Lovibond & Lovibond, 1995) is used. The DASS is a 42-item self-report instrument with 3 sub-scales. Each scale comprises 14 items assessing the negative emotional states of depression, anxiety and stress.
Change in Stress | 3, 5, and 6 months
  The Depression Anxiety Stress Scale - DASS (Lovibond & Lovibond, 1995) is used. The DASS is a 42-item self-report instrument with 3 sub-scales. Each scale comprises 14 items assessing the negative emotional states of depression, anxiety and stress.